CLINICAL TRIAL: NCT03619356
Title: Investigation of Hemoglobin Oxygenation With Third Harmonic Generation Microscopy
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201709032RINB
Record Dates: First submitted 2018-06-11; First posted 2018-08-07 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2023-11

CONDITIONS: Hypoxia; Oxygen Deficiency; Tumor; Diabetes
Keywords: hemoglobin; oxygenation concentration; tumor; diabetes
MeSH Terms: conditions — Hypoxia; Neoplasms; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The specific aims of the project are performing a pre-clinical study on a human model and evaluating the oxygenation and other status of human erythrocytes by spectrally-resolved third harmonic generation (srTHG) microscopy . By analyzing the partitioned third harmonic generation (THG) spectra of oxygenated and deoxygenated erythrocytes ex vivo, the investigators aim to provide a reference standard for quantifying oxygenation and molecular status in this project.

DETAILED DESCRIPTION:
Recently, oximeter, detecting the spectral response at wavelengths of 660nm and 940nm, is widely used to measured oxygenation status. Its low spatial resolution and limited penetration depth in human skin, however, restrict the oximeter in clinical application especially for early detection of cancer. In early-stage cancer development, angiogenesis and oxygen depletion around tumor are two important indicators of tumor growth. If an angiogenesis and low oxygenation status can be identified simultaneously, the investigators can point out the early-stage tumor from normal tissue easily.

The investigators have been working towards the development of third harmonic generation microscopy systems and reported the success of revealing morphology in human skin specimen. Since THG process is based on virtual transition without energy deposition, THG microscopy enables imaging ex vivo specimens without extra label and invasive procedure. To further investigate biological process of biomaterials, the investigators develop a srTHGM where THG spectrum is partitioned to analyze during imaging process. In this project, the investigators aim to elucidate oxygenation concentration and other specific biological molecular of red blood cells through the srTHG microscopy system.

The abilities to reveal structure morphology and its corresponding biological information in situ would provide assistance to diagnose early-stage of tumor and other diseases as well as a potential support in clinical treatment.

ELIGIBILITY:
Inclusion Criteria:

* older than 20 years old

Exclusion Criteria:

* Vulnerable groups, such as pregnant women, prisoners, students, mentally handicapped, aborigines, etc.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Volunteers with any genders with the age older than 20 years.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-02-05 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Observe the extent of tumor growth via morphological information | 2 years
  To observe the extent of tumor growth (with units of mm2) via morphological information. Morphological information are presented as density and shape of red blood cells.
Observe the extent of tumor growth via spectral THG intensity distribution | 2 years
  To observe the extent of tumor growth (with units of mm2) via spectral THG distributions. The spectral distributions are presented by the ratio between different channels. And the ratio can be calculated by analyzing the excited fluorescence intensity.
Change in spectral THG strength distribution | 2 years
  Obtain THG strength in 3 different channels for chemically treated whole blood samples for oxygenation, deoxygenation and other status. The spectral distributions are presented by the ratio between different channels.

SECONDARY OUTCOMES:
Quantify the extent of diseases in spectral THG strength distribution | 1 year
  With calculating the ratio of THG strength for chemically treated whole blood samples for oxygenation and deoxygenation and other status from different channels, the extent of other diseases can be quantified.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan